CLINICAL TRIAL: NCT02386423
Title: Efficacy and Safety of the RESTIFFIC™ Brand Pressure Application System, the Restless Leg Relaxer to Reduce the Symptoms of Moderate to Severe Restless Leg Syndrome
Brief Title: RESTIFFIC™ Foot Wrap Reduces Moderate to Severe Restless Leg Syndrome
Acronym: RESTIFFIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sorg1
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Restless Leg Syndrome
Keywords: RLS; Willis-Ekbom
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RESTIFFIC (Experimental): RESTIFFIC™ Brand Pressure Application System
  Interventions: Device: RESTIFFIC™ Brand Pressure Application System

INTERVENTIONS:
Device: RESTIFFIC™ Brand Pressure Application System — The device, RESTIFFIC™, was administered intermittently through the course of the study: one-week baseline period without the device (days 1-7), three weeks of initial testing with the device (days 8-28), a subsequent one-week period without the device (days 29-35), and three weeks of subsequent testing with the device (days 36-56).
  Other Names: Restless Leg Relaxer

SUMMARY:
The purpose of this study is to determine the safety and efficacy of RESTIFFIC™, a foot wrap that produces adjustable targeted pressure on specific muscles in the feet, to reduce the symptoms of moderate to severe primary Restless Legs Syndrome.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS), or Willis-Ekbom Disease, is a neurologic disorder causing unpleasant sensations and an urge to move the legs when the person is at rest. The sensations are relieved by movement. Loss of sleep associated with RLS can cause extreme fatigue, affecting concentration, which may produce anxiety and depression, resulting in a poor quality of life. Prevalence in the general population is 5% to 10%. In approximately 3%, symptoms are so severe that treatment is sought. Potent drugs, such as opioids, central nervous system depressants, anticonvulsants, and dopamine agonists have been used to ease symptoms, each with several side effects.

Anecdotal evidence suggested that pressure on specific foot muscles decreases symptoms of moderate to severe primary restless legs syndrome. In the RESTIFFIC™ study, patients served as their own negative controls, wearing the RESTIFFIC™ devices intermittently, while completing surveys related to RLS throughout the study. Physicians also completed surveys related to quality of life. Meta-analysis was used to compare RESTIFFIC™ to historic reports of ropinirole and placebo pill. Demographics, disease severity,inclusion/exclusion criteria, assessment tools were similar among studies.

ELIGIBILITY:
Inclusion Criteria:

Otherwise healthy adults between the ages of 18 and 75 years who were diagnosed with moderate to severe RLS were recruited from Erie and the surrounding regions. The patient was examined by the physician and screened using the medical history, the International RLS study group diagnostic criteria, and International RLS Study (IRLSS) Rating Scale.

To be included, patients had to have: (1) a total score of 15 or greater on the International RLS Rating Scale; (2) evening and nighttime symptoms with sleep impairment (by self-report) due to RLS; and (3) RLS for at least six months with symptoms at least two to three times per week. The potential was for at least 12 and as many as 42 episodes of RLS during the treatment period.

Exclusion Criteria:

The patient was excluded if he/she had any serious medical conditions or conditions that may have presented a safety concern or that may have impacted efficacy assessment, eg, taking drugs like antidepressants known to affect RLS. Medical conditions included, but were not limited to: claudication, nerve problems, fragile, thin skin, impaired wound healing; poor circulation, injury to feet or legs, movement problems, inability to sit still or remain motionless, involuntary movements similar to a tic, sleep disorders, parasomnias involving abnormal movements, narcolepsy, obstructive sleep apnea, nighttime discomfort not due to RLS, secondary RLS, or Parkinson's Disease. Patients on drug treatment for RLS must have been discontinued treatment for at least 30 days. (Note: None of our patients were on drug treatment for RLS.) Through history and physical examination, the physician distinguished RLS from other disorders such as periodic Limb Movement Disorder (footnote 5)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in International Restless Legs Syndrome Study Rating Scale | Change in International RLS Study Group (IRLSS) Rating Scale from baseline to Day 56 Study end

SECONDARY OUTCOMES:
Clinical Global Impression Scale | Four CGI Scales, one each on Days, 1, 29, 36, and 57

OTHER OUTCOMES:
Meta-analysis used to compare change in IRLSS scores in RESTIFFIC to change in IRLSS scores for ropinirole and placebo pill (historic reports) | Baseline to end of study
Number and type of adverse events as a measure of safety and tolerability of RESTIFFIC™ vs ropinirol and placebo (historic reports) | Baseline to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis J Kuhn, PhD, Study Director — Lake Erie Research Institute; Daniel J Olson, DPM, AACFAS, Principal Investigator — Baycity Associates in Podiatry Inc
Locations (1):
- Baycity Associated in Podiatry Inc, Erie, Pennsylvania, United States

REFERENCES:
- [Background] Bogan RK, Fry JM, Schmidt MH, Carson SW, Ritchie SY; TREAT RLS US Study Group. Ropinirole in the treatment of patients with restless legs syndrome: a US-based randomized, double-blind, placebo-controlled clinical trial. Mayo Clin Proc. 2006 Jan;81(1):17-27. doi: 10.4065/81.1.17. PMID 16438474
- [Background] Trenkwalder C, Garcia-Borreguero D, Montagna P, Lainey E, de Weerd AW, Tidswell P, Saletu-Zyhlarz G, Telstad W, Ferini-Strambi L; Therapy with Ropiunirole; Efficacy and Tolerability in RLS 1 Study Group. Ropinirole in the treatment of restless legs syndrome: results from the TREAT RLS 1 study, a 12 week, randomised, placebo controlled study in 10 European countries. J Neurol Neurosurg Psychiatry. 2004 Jan;75(1):92-7. PMID 14707315
- [Background] Walters AS, Ondo WG, Dreykluft T, Grunstein R, Lee D, Sethi K; TREAT RLS 2 (Therapy with Ropinirole: Efficacy And Tolerability in RLS 2) Study Group. Ropinirole is effective in the treatment of restless legs syndrome. TREAT RLS 2: a 12-week, double-blind, randomized, parallel-group, placebo-controlled study. Mov Disord. 2004 Dec;19(12):1414-23. doi: 10.1002/mds.20257. PMID 15390050
- [Derived] Kuhn PJ, Olson DJ, Sullivan JP. Targeted Pressure on Abductor Hallucis and Flexor Hallucis Brevis Muscles to Manage Moderate to Severe Primary Restless Legs Syndrome. J Am Osteopath Assoc. 2016 Jul 1;116(7):440-50. doi: 10.7556/jaoa.2016.088. PMID 27367949